CLINICAL TRIAL: NCT05867914
Title: A Within-subject Device-setting Escalation Early Feasibility Study Evaluating the Safety, Tolerability, and Functionality of 3P-100 in Subjects With PH-ILD
Brief Title: Early Feasibility Study Evaluating the 3P-100 Device in Subjects With PH-ILD
Acronym: EFS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Pole Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3P-100-ILD-00
Record Dates: First submitted 2023-05-01; First posted 2023-05-22 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Hypertension, Pulmonary; Lung Diseases, Interstitial
Keywords: inhaled NO, PH-ILD
MeSH Terms: conditions — Hypertension, Pulmonary; Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: eNOfit system delivering iNO
Masking Description: eNOfit an Electric Nitric Oxide (NO) Ambulatory Production and Delivery System, Delivering Nitric Oxide for Inhalation
  The treatment period with inhaled Nitric Oxide (iNO) will include start of iNO at a device setting of 2 mg/hr iNO for 2 hours (+15 minutes), device setting escalation to 6 mg/hr iNO for 2 hours (+15 minutes) and then weaning of iNO treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Inhaled Nitric Oxide (iNO) (Experimental): eNOfit an Electric Nitric Oxide (NO) Ambulatory Production and Delivery System, Delivering Nitric Oxide for Inhalation
  The treatment period with inhaled Nitric Oxide (iNO) will include start of iNO at a device setting of 2 mg/hr iNO for 2 hours (+15 minutes), device setting escalation to 6 mg/hr iNO for 2 hours (+15 minutes) and then weaning of iNO treatment
  Interventions: Device: Inhaled Nitric Oxide (iNO)

INTERVENTIONS:
Device: Inhaled Nitric Oxide (iNO) — eNOfit system delivering iNO

SUMMARY:
A trial to evaluate the safety, tolerability, and functionality of 3P-100, in subjects with Pulmonary Hypertension (PH) accompanying Interstitial Lung Disease (ILD), PH-ILD

DETAILED DESCRIPTION:
This is a multi-center early feasibility study evaluating the safety and tolerability of the 3P-100 device which creates and delivers iNO (2 mg/hr and 6 mg/hr) for the treatment of subjects with PH-ILD. All subjects will use the 3P-100 device and receive iNO (2 mg/hr and 6 mg/hr) via the 3P-100 device, aiming for ~4-4.5 hours of treatment across both device settings.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 22 to < 85 years old
2. Provides signed informed consent for study participation
3. Diagnosis of any form of advanced Interstitial Lung Disease or Combined Pulmonary Fibrosis and Emphysema (CPFE) at any time, based on clinical, pulmonary function, serological, and Computed Tomography (CT) radiologic evidence (which demonstrates evidence of moderate to severe diffuse parenchymal lung disease)
4. A prior Right Heart Catheterization (RHC) at any time before SV that demonstrates PH with a Pulmonary Vascular Resistance (PVR) >2.0 Wood Units (WU), a mean Pulmonary Arterial Pressure (mPAP) > 20 mmHg, and a Pulmonary Capillary Wedge Pressure (PCWP) ≤ 15 mmHg. A PCWP >15 mmHg is not exclusionary if a left ventricular end diastolic pressure (LVEDP) is available and is ≤ 15 mmHg by left heart catheterization AND/OR Previous Echocardiography with an intermediate/high probability of PH (European Society of Cardiology definition)
5. New York Heart Association (NYHA) functional class II-IV
6. Self-reported use of long-term O2 therapy (LTOT) less than or equal to 10 L/minute at rest and while exercising, defined as use for at least 12 hours per day for at least 30 days prior to SV
7. Is willing to comply with treatment with iNO and procedures including using the 3P-100 device and wearing a nasal cannula for at least 4 hours at V1
8. Is able to wear a 3P-100 device while sitting and ambulating intermittently in the clinic area for at least 30 minutes during SV
9. Women of child-bearing potential must agree to use the methods of birth control indicated in Appendix 1 from consent through the Telephone Call at V1 +1 Day

Exclusion Criteria:

1. History or diagnosis by Investigator evaluation during SV of World Health Organization (WHO) Group I, II, IV, or V PH
2. NYHA class IV patients who are medically unfit to participate i.e., are constantly breathless at rest or have frequent symptoms of chest pain or syncope at rest or with activity
3. History or diagnosis of acute or chronic left heart failure at any time as evidenced by one or more of the following:

   1. PCWP > 15 mmHg on a previous RHC (unless LVEDP is ≤15 mmHg) AND/OR LVEDP >15 mmHg by left heart catheterization
   2. Previous echocardiographic findings of left ventricular systolic dysfunction with ejection fraction < 40%
   3. Cardiogenic pulmonary edema
   4. History of left heart failure (Prior or current use of medications given solely for the treatment of systemic hypertension are allowed)
4. History of hereditary methemoglobinemia
5. History of the following cardiovascular conditions:

   1. Stenting or Coronary Artery Bypass Graft (CABG) within 60 days prior to SV
   2. Myocardial infarction within the 60 days prior to SV
   3. Unstable angina pectoris in the 60 days prior to SV
   4. Intermittent atrial fibrillation, supraventricular tachycardia, and serious ventricular arrhythmias (e.g., ventricular tachycardia) within 60 days prior to SV. Ablated atrial flutter or Wolf-Parkinson-White (WPW) bypass tract conduction are not exclusionary
   5. Cerebrovascular accident within the 60 days prior to SV
6. Has within 30 days prior to SV or during the Screening period

   1. Participated in any clinical study involving an investigational drug, investigational biologic, or investigational device
   2. Required unplanned hospitalization for any reason
   3. Had an exacerbation of ILD requiring administration of oral or parenteral antibiotic
7. Has within the 30 days prior to SV or during the Screening period required initiation or changes in the regimen (including agents, dose, and frequency) of medications prescribed for the treatment of ILD, including but not limited to immunosuppressive / immunomodulatory medications, systemic oral or parenteral corticosteroids, and monoclonal antibodies
8. Has within 30 days prior to SV, or any time during Screening period taken one or more of the following medications or supplements chronically:

   1. Oral, inhaled, or parenteral medications for the treatment of Pulmonary Arterial Hypertension (PAH) irrespective of the route of administration including, but not limited to,

      * high dose calcium channel blockers
      * riociguat
      * prostacyclins
      * prostacyclin analogues
      * prostacyclin receptor agonists (e.g., selexipag)
      * phosphodiesterase type 5 (PDE5) inhibitors (e.g., sildenafil) if the subject is on inhaled treprostinil
      * endothelin receptor antagonists
   2. Inhaled treprostinil (approved for PH-ILD), if the subject is on a PDE5 inhibitor for PH-ILD

      Note: Inhaled treprostinil is not exclusionary as a monotherapy, however, the concurrent use of both a PDE5 inhibitor (e.g., sildenafil) and inhaled treprostinil is exclusionary. The use of either a PDE5 inhibitor or inhaled treprostinil will be allowed if both conditions are met:
      * The PDE5 inhibitor or inhaled treprostinil was started more than 30 days prior to the SV.
      * There have been no changes in the PDE5 inhibitor or inhaled treprostinil dosage within 30 days prior to the SV.
   3. Nitrates, regardless of route of administration
   4. Supplements containing L-arginine
   5. Agents or medications capable of inducing methemoglobinemia where any of the SV/V1 metHb average measurements via co-oximeter are > 3.5%

   Subjects should not be weaned from these therapies for the purpose of enrollment.
9. Is breastfeeding or lactating at the time of SV or intends to breastfeed at any time during their participation in the study
10. Has one of the following in their medical record or through testing performed:

    1. Positive urine pregnancy test at SV or on V1 (results of the test are to be known prior to initiation of the iNO)
    2. Hemoglobin < 10 g/dL (100 g/L) within 30 days of SV
    3. HbA1c > 10% within 30 days of SV
    4. Glomerular Filtration Rate (GFR) < 30 mL/min/1.73 m2 , calculated using the Creatinine Clearance (CKD-EPI) calculation method within 30 days of SV
    5. Methemoglobin > 3.5% at SV or V1 via co-oximeter measurements
    6. Thrombocytopenia with a platelet count < 50 x 103 /µL (< 50 X 109/L) within 30 days of SV
11. Has any condition at SV/V1 that could constitute a safety concern during participation in the study or could interfere with the subject's ability to comply with adherence to iNO, including but not limited to:

    1. Uncontrolled systemic hypertension defined by systolic Blood Pressure (BP) > 180 mmHg and/or a diastolic BP > 110 mmHg measured manually after 20 minutes at rest on prescribed resting O2
    2. History of alcohol or substance abuse within the past 365 days prior to SV. Drugs documented as prescribed by a physician or use of edible marijuana if legal in the state of residence may be allowed with approval of the Medical Monitor. Smoking and vaping of any substance is prohibited (e.g., nicotine or marijuana)
    3. History of poor compliance with prior clinical studies
    4. Acute or chronic physical impairment (other than dyspnea due to ILD) (e.g., neurologic, musculoskeletal, or orthopedic disorder, or dependence on mobility aids such as a cane or walker) that would limit the ability to carry and operate the 3P-100 device together with their O2 system
    5. Severe right heart failure confirmed by the investigator as evidenced by two or more of the following: elevated jugular venous pressure, peripheral edema, hepatic congestion and/or ascites
    6. Other known coagulopathies
12. Is a relative of Third Pole, the Contract Research Organization (CRO) or other vendor, or investigational site/institutional personnel
13. Has during the SV one or more of the following results:

    1. Forced Expiratory Volume (FEV1)/Forced Vital Capacity (FVC) ratio < 0.7 except for CPFE
    2. FVC < 40% predicted

Ages: 22 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-03-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events [By evaluating safety and tolerability of ascending device settings of iNO administered in the clinic with the 3P-100 device in PH-ILD] | Day 1
  Incidence of Adverse Events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Effect of iNO on oxygen saturation | Day 0
  Assessment of the effect of iNO on oxygen saturation as assessed by SpO2 (Pulse Oximetry)
Device Usability Questionnaire (Created by Third Pole) | Day 0
  Assessment of the responses on the Device Usability Questionnaire completed by the Subject.
  It is a 5 point scale.
  1 = Very Difficult, Completely Unacceptable 5 = Very Easy, Completely Acceptable

CONTACTS AND LOCATIONS:
Overall Officials: Philip Silkoff, MD, Study Director — Chief Medical Officer
Locations (3):
- United States (3):
  - TGH/USF Center for Advanced Lung Disease and Lung Transplant, Tampa, Florida
  - University of Cincinnati, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No